CLINICAL TRIAL: NCT01599195
Title: Use of Amplified Sound Signal to Identify Presence of Carotid and Femoral Stenosis
Status: Terminated | Type: Observational
Why Stopped: Enrollment did not progress as anticipated
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Jonathan Dissin, MD, Principal Investigator, Albert Einstein Healthcare Network
Other Study IDs: HN 4209
Record Dates: First submitted 2012-05-02; First posted 2012-05-15 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Carotid Stenosis; Femoral Arterial Stenosis; Carotid Bruit Asymptomatic; Carotid Murmur
Keywords: carotid stenosis; femoral artery ischemia; carotid bruit asymptomatic; carotid murmur
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- adults: adults audiodoc use to evaluate for carotid or femoral bruit
  Interventions: Device: AudioDoc

INTERVENTIONS:
Device: AudioDoc — AudioDoc will be used to identify the carotid and femoral bruit

SUMMARY:
The purpose of the study is to test a new amplified stethoscope(AudioDoc) that can detect the presence of bruit by using an acoustic signal to represent the bruit. This pilot study will address two questions: is there a detectable difference in recorded sound signal of carotid and femoral bruit when compared to sound signals captured when there is no bruit present; is the use of a visual recorded signal more accurate in identifying carotid and femoral bruit when compared to traditional auscultation with a regular stethoscope and ultrasound.

DETAILED DESCRIPTION:
Recorded signals are stored on a laptop computer. The signals later undergo Fourier analysis are then compared to the findings on carotid ultrasoud as to degree of stenosis. Subjects with high grade stenosis in which no bruit was ascultated but in which carotid ultrasound data suggests a bruit may be present are studied for soft /inaudible bruits. When available, data will be correlated to CT/conventional angiographic studies.

ELIGIBILITY:
Inclusion Criteria:

* age 19-90 years
* having clinical ultrasound evaluation of carotid or femoral artery

Exclusion Criteria:

* under age 19; over age 90 years

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: any person age 19 through 90 years who have been clinically determined to require evaluation of carotid or femoral arteries for suspected stenosis
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Comparison of bruit signal obtained from the amplified stethoscope(AudioDoc) to that found by conventional ultrasonography. | subjects will be followed for duration of hospital stay, typically four days.

SECONDARY OUTCOMES:
To assess the frequency spectral differences obtained from the different recording modalities | duration of hospital stay, typically four days

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dissin, MD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Albert Einstein Healthcare Network, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No